CLINICAL TRIAL: NCT02817152
Title: Low-level Laser Therapy in the Treatment of Chronic Periodontitis in Type 2 Diabetics: Split-mouth Double-blind Randomized Clinical Trial
Brief Title: Low-level Laser Therapy in the Treatment of Chronic Periodontitis in Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Nídia Cristina Castro dos Santos, DDS, MS, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NCSlaser
Record Dates: First submitted 2016-06-10; First posted 2016-06-29 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Periodontitis; Diabetes Mellitus
Keywords: periodontal treatment; low-level light therapy
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus | interventions — Periodontal Debridement; Debridement; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Periodontal ultrasonic debridement (Sham Comparator): Periodontal pockets received ultrasonic periodontal debridement intervention.
  Interventions: Procedure: Periodontal ultrasonic debridement
- Low-level laser therapy (Active Comparator): Periodontal pockets received ultrasonic periodontal debridement plus low-level laser therapy intervention.
  Interventions: Procedure: Periodontal ultrasonic debridement; Device: Debridement plus low-level laser therapy

INTERVENTIONS:
Procedure: Periodontal ultrasonic debridement — Periodontal pockets received periodontal ultrasonic debridement intervention.
  Other Names: periodontal debridement; ultrasonic debridement
Device: Debridement plus low-level laser therapy — Ultrasonic debridement plus low-level laser therapy.
  Other Names: low-level light therapy; low-power laser therapy; low-intensity laser therapy
  Arms: Low-level laser therapy

SUMMARY:
The aim of this study was to investigate the local effect of adjunct low-level laser therapy (LLLT) for the treatment of moderate to severe chronic periodontitis in type 2 diabetic patients.

DETAILED DESCRIPTION:
The aim of this study was to investigate the local effect of adjunct low-level laser therapy (LLLT) for the treatment of moderate to severe chronic periodontitis in type 2 diabetic patients. Twenty poorly-controlled type 2 diabetic patients with moderate to severe generalized chronic periodontitis were selected. Two periodontal pockets with Probing Depth (PD) and Clinical Attachment Level (CAL) ≥ 5mm received ultrasonic periodontal debridement (UPD) only (control group) or UPD with LLLT (test group). Clinical measures, such as PD, CAL, Gingival Recession (GR), Bleeding on Probing (BoP), and Plaque Index (PI), were collected and compared at baseline, 30, 90, and 180 days. The adjunct application of LLLT to UPD had no additional benefits for PD reduction and CAL gain, meaning that both investigated therapies were efficient for the treatment of chronic periodontitis in type 2 diabetics. Nevertheless, additional LLLT application showed better results for GR then UPD only.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 35; diagnosis of type 2 diabetes for ≥ 5 years; diabetes treatment with oral hypoglycemic agents or insulin supplementation and diet; glycated hemoglobin (HbA1c) levels from 6.5% to 11%; at least 15 teeth (excluding third molars and teeth indicated for extraction); and moderate to severe generalized chronic periodontitis.

Exclusion Criteria:

* The exclusion criteria were: medical conditions that required prophylactic antimicrobial coverage; periodontal mechanical therapy in the previous 6 months; antimicrobial therapies in the previous 6 months; anti-inflammatory therapies in the previous 6 months; systemic conditions other than diabetes that could affect the progression of chronic periodontitis; current use of medication that could interfere with periodontal response to treatment; pregnancy or lactation; and smoking.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Probing depth change from baseline to 30, 90, and 180 days through periodontal probing | baseline, 30 days, 90 days, 180 days

SECONDARY OUTCOMES:
Clinical attachment level change from baseline to 30, 90, and 180 days through periodontal probing | baseline, 30 days, 90 days, 180 days
Gingival recession change from baseline to 30, 90, and 180 days through periodontal probing | baseline, 30 days, 90 days, 180 days
Bleeding on probing change from baseline to 30, 90, and 180 days through periodontal probing | baseline, 30 days, 90 days, 180 days
Plaque index change from baseline to 30, 90, and 180 days through periodontal probing | baseline, 30 days, 90 days, 180 days

OTHER OUTCOMES:
Glycated hemoglobin | Baseline, 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, DDS, MS, PhD, Study Director — UPECLIN HC FM Botucatu Unesp

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aykol G, Baser U, Maden I, Kazak Z, Onan U, Tanrikulu-Kucuk S, Ademoglu E, Issever H, Yalcin F. The effect of low-level laser therapy as an adjunct to non-surgical periodontal treatment. J Periodontol. 2011 Mar;82(3):481-8. doi: 10.1902/jop.2010.100195. Epub 2010 Oct 8. PMID 20932157